CLINICAL TRIAL: NCT00610285
Title: A Feasibility Study of Image Guided Noninvasive Single Fraction Stereotactic Radiosurgery for the Treatment of Brain Metastases
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-110
Record Dates: First submitted 2008-01-14; First posted 2008-02-07 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Brain Cancer
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- non-invasive immobilization system: This is a feasibility study to evaluate the accuracy of an alternative, non-invasive immobilization system in combination with image guided patient setup for SRS treatments. The aim is to determine whether or not the non-invasive system can provide comparable accuracy as the conventional invasive head ring system. If successful, patient discomfort can be significantly reduced for such treatments.
  Interventions: Other: Fabrication of thermoplastic face (The Orfit thermoplastic face mask system is routinely used for the treatment of brain and head)

INTERVENTIONS:
Other: Fabrication of thermoplastic face (The Orfit thermoplastic face mask system is routinely used for the treatment of brain and head) — Each patient in the protocol will receive their regularly scheduled SRS treatment plus an additional mock treatment using the non-invasive immobilization system.

SUMMARY:
Stereotactic radiosurgery (SRS) is a way to accurately treat brain tumors. SRS involves the use of a special head frame to keep the head from moving during treatment. The head frame makes very accurate treatment possible. The frame must be attached to the skull with special pins. It feels very tight and can hurt. A special immobilization device can be used to keep the head from moving.

This device does not need any pins and does not hurt. We would like to see if the new way of holding the head still can be used for SRS. This is the purpose of the study. New X-Ray machines can be used to find if the head has moved in the mask. We hope that we can use these new tools to treat brain tumors just as accurately without using a head frame. It will make treatment more comfortable for the patient. This is why we are asking patients to join the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy with the presence of intraparenchymal brain metastases.
* A diagnostic contrast enhanced MRI demonstrating the presence of brain metastases performed within two weeks prior to registration.
* Age ≥ 18 years.
* Must be scheduled or planning to be scheduled for SRS treatment.
* Karnofsky performance status ≥60.
* Patient must sign a study-specific informed consent form. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the patient's legal representative.

Exclusion Criteria:

* Unable to provide informed consent
* Major medical illness including poor cardiac or pulmonary status which would result in inability of the patient to lie down for the procedure.
* Inability to obtain histologic proof of malignancy.
* Younger than 18 years of age.
* Serum creatinine > 1.3 mg/dl.
* Karnofsky performance status of ≤50.
* Allergy to either CT or MR contrast dyes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC Clinic
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2005-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Use the kilovoltage On-Board Imager (kVOBI) to precisely measure the setup accuracy of conventional, invasive frame SRS on 10 patients | conclusion of study

SECONDARY OUTCOMES:
Use the kilovoltage On-Board Imager (kVOBI) to precisely measure the accuracy of an image guided non-invasive (Aktina stereotactic localizer) immobilization system on the same 10 patients as in above. | conclusion of study
Compare setup accuracy of both systems above, and investigate the feasibility of 'system B' as replacement for 'system A' for single fraction SRS | conclusion of the study
Compute mean and standard deviation of the intra-fractional motion for non-invasive SRS. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org